CLINICAL TRIAL: NCT03939702
Title: Pharmacokinetic and Metabolism of [14^C] BMS-986177 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CV010-036
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-08

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-Bile Collection (Active Comparator): On Day 1, all participants will receive a single oral solution dose of 200 mg [14C] BMS-986177 containing approximately 88 micro Ci of total radioactivity (TRA). Participants will remain in the clinical facility until at least Day 7 and will be discharged when release criteria are met or until Day 12
  Interventions: Drug: BMS-986177
- Bile Collection (Active Comparator): On Day 1, all participants will receive a single oral solution dose of 200 mg [14C] BMS-986177 containing approximately 88 micro Ci of total radioactivity (TRA). Approximately 1 hour after study drug administration, an ND tube may be positioned in approximately 3 selected participants for collection of bile.Participants will remain in the clinical facility until at least Day 7 and will be discharged when release criteria are met or until Day 12
  Interventions: Drug: BMS-986177

INTERVENTIONS:
Drug: BMS-986177 — An orally administered anticoagulant to prevent and treat thromboembolic events

SUMMARY:
This is an ADME study. Human radiolabeled mass balance studies are performed as part of drug development to obtain information about the absorption, distribution, metabolism, and excretion (ADME) of a study treatment. The goals of human ADME studies include the assessment of absorption, distribution, routes and rates of excretion, mass balance, and metabolite profile and identification.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF
* Healthy Male
* Body mass index of 18.0 to 32.0 kg/m2, inclusive.
* Agreement to use approved contraception for 94 days post treatment
* Agreement to not donate sperm for 94 days post treatment

Exclusion Criteria:

* Acute or chronic illness
* GI disease current or recent
* History of dizziness or recurring headaches
* Head injury within last 2 years
* GI surgery
* History or evidence of abnormal bleeding

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Born male
Enrollment: 9 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Assess PK Cmax of a dose of [14C]BMS-986177 | Day 1-12
  Cmax
Assess PK AUC(INF) of a dose of [14C]BMS-986177 | Day 1-12
  AUC(INF)
Assess PK AUC(0-T) of a dose of [14C]BMS-986177 | Day 1-12
  AUC(0-T)
Assess PK Tmax of a dose of [14C]BMS-986177 | Day 1-12
  Tmax
Assess PK T-HALF of a dose of [14C]BMS-986177 | Day 1-12
  T-HALF
Assess PK CL/F of a dose of [14C]BMS-986177 | Day 1-12
Assess PK Vz/F of a dose of [14C]BMS-986177 | Day 1-12
  Vz/F
Assess PK AUC of a dose of [14C]BMS-986177 | Day 1-12
  AUC(BMS-986177)
Assess PK AUC(TRA) of a dose of [14C]BMS-986177 | Day 1-12
  AUC(TRA)
Assess PK Plasma AUC(TRA) of a dose of [14C]BMS-986177 | Day 1-12
  Plasma AUC(TRA)
Assess PK Blood AUC(TRA) of a dose of [14C]BMS-986177 | Day 1-12
  Blood AUC(TRA)
Assess the CLR of [14C]BMS-986177 | Day 1-12
  CLR
Assess the %UR of [14C]BMS-986177 | Day 1-12
  %UR
Assess the %FE of [14C]BMS-986177 | Day 1-12
  %FE
Assess the %BE of [14C]BMS-986177 | Day 1-12
  %BE (if applicable)
Assess the %Total recovery of [14C]BMS-986177 | Day 1-12
  %Total recovery

SECONDARY OUTCOMES:
Asess the Incidence of AEs of a single oral dose of 200 mg [14C] BMS-986177 | Day 1-12
  Incidence of AEs
Asess the Incidence of SAEs of a single oral dose of 200 mg [14C] BMS-986177 | Day 1-12
  Incidence of SAEs
Asess the Incidence of AEs leading to discontinuation of a single oral dose of 200 mg [14C] BMS-986177 | Day 1-12
  Incidence of AEs leading to discontinuation
Assess the vital signs of a subject dosed with single oral dose of 200 mg [14C] BMS-986177 | Day 1-12
  results of vital sign examination
Assess the ECGs of subjects dosed with single oral dose of 200 mg [14C] BMS-986177 | Day 1-12
  ECG physical examinations
Assess the clinical lab tests of a single oral dose of 200 mg [14C] BMS-986177 | Day 1-12
  Results of Clinical laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States